CLINICAL TRIAL: NCT03402828
Title: Body PSOriasis: Long-term Relapse Control in Patients With Psoriasis Vulgaris in Daily Clinical Practice of Russian Dermatologists.
Brief Title: Body PSOriasis: Long-term Relapse CONTROL
Acronym: PSO-CONTROL
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-PSORIASIS-1379
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2019-12

CONDITIONS: Psoriasis Vulgaris
Keywords: Topicals; Long-term

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Any topical drug treatment — Any treatment strategy used to prevent relapse of psoriasis symptoms
  Other Names: Non-drug topicals

SUMMARY:
This non-interventional study of real-life clinical practice strategies for long-term relapse control in patients with psoriasis vulgaris is planned to enroll 650 adult patients from 60-100 Russian dermatology sites and follow the patients for up to 52 weeks. The study will map actual strategies and focus on patients' and dermatologists' experience with the different topicals used, including unspecified products with and without active drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned to receive topical treatment of any kind to prevent relapse of symptoms
* Written informed consent

Exclusion Criteria:

* Contraindications to selected treatment
* Ongoing systemic treatment of psoriasis with steroids, anti-inflammatory drugs or phototherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with psoriasis vulgaris attending one of the participating outpatient dermatology clinics entering a phase of prevention of relapse of psoriasis symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 764 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Time of relapse | Up to 52 weeks
  Length of relapse free period after start of maintenance strategy

SECONDARY OUTCOMES:
Dermatology Life Quality Index | Up to 52 weeks
  Standard QoL measure within dermatology
PGA (physician's global assessment of symptoms) | Up to 52 weeks
  5-point verbal rating scale
PsGA (patient's global assessment of symptoms) | Up to 52 weeks
  5-point verbal rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Petrunin, MD PhD, Study Director — Leo Pharmaceutical Products LLC
Locations (1):
- The State Autonomous Foundation of Public Health "Republic Clinical Dermatovenereological Dispensary" of the Republic of Tatarstan, Kazan', Tatarstan Republic, Russia

IPD SHARING:
Plan to Share IPD: No